CLINICAL TRIAL: NCT00439738
Title: A 16-week Double-blind, Randomized, Multicenter, Force-titration Study to Evaluate the Antihypertensive Efficacy of Valsartan/Hydrochlorothiazide (HCTZ) Therapy Compared to HCTZ Based Therapy in Obese, Hypertensive Patients
Brief Title: Safety/Efficacy of Valsartan/Hydrochlorothiazide Combination Compared to Hydrochlorothiazide in Obese Hypertensive Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631BUS06
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2009-02-10 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
Keywords: Obesity, hypertension, valsartan/hydrochlorothiazide
MeSH Terms: conditions — Hypertension; Obesity | interventions — Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- valsartan/HCTZ (Experimental)
  Interventions: Drug: Valsartan/HCTZ
- HCTZ +Amlodipine (Active Comparator)
  Interventions: Drug: HCTZ + Amlodipine

INTERVENTIONS:
Drug: HCTZ + Amlodipine — * 12.5 mg HCTZ capsules
  * 25 mg HCTZ capsules
  * 5 mg amlodipine capsules
  * 10 mg amlodipine capsules
  Arms: HCTZ +Amlodipine
Drug: Valsartan/HCTZ — * 160 mg film-coated valsartan tablets
  * 320 mg film-coated valsartan tablets
  * 12.5 mg HCTZ capsules
  * 25 mg HCTZ capsules
  Arms: valsartan/HCTZ

SUMMARY:
The purpose of this study is to compare the blood pressure lowering efficacy of valsartan/hydrochlorothiazide (HCTZ) compared to hydrochlorothiazide for the treatment of obese hypertensive (mean sitting systolic blood pressure [MSSBP] >150 mmHg) patients.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Moderate or severe high blood pressure defined as systolic blood pressure (the top number) greater than or equal to 150 mmHg and diastolic blood pressure (the bottom number) less then 110 mmHg
* Central (abdominal) obesity

Exclusion Criteria:

* Systolic blood pressure (the top number) greater than or equal to 180 mmHg and diastolic blood pressure (the bottom number) greater than or equal to 110 mmHg
* Currently taking more then 3 medications to treat high blood pressure
* Inability to stop all current blood pressure medications if any up to 4 weeks
* History of Type 1 or Type 2 diabetes
* History of stroke, mini-stroke (transient ischemic attack) or heart attack within the last 6 months
* History of or current diagnosis of congestive heart failure
* History of cancer within the past 5 years with the exception of localized basal cell carcinoma or squamous cell carcinoma
* Women who are pregnant or nursing
* Alcohol or drug abuse within the last 2 years

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Terence T. Hart, MD, Muscle Shoals, Alabama
  - Westlake Medical Research, Westlake Village, California
  - Oklahoma Cardiovascular & Hypertension, Oklahoma City, Oklahoma
  - Northeast Tarrant Internal Medicine Assoc, Euless, Texas
  - Frandsen Family Medicine, Port Orchard, Washington

REFERENCES:
- [Derived] Deedwania PC, Zappe DH, Egan BM, Purkayastha D, Samuel R, Sowers JR. Does response of RAS blockade on serum K+ levels influence its glycemic-mitigating response when combined with hydrochlorothiazide? J Clin Hypertens (Greenwich). 2012 Jul;14(7):415-21. doi: 10.1111/j.1751-7176.2012.00635.x. Epub 2012 Apr 26. PMID 22747613
- [Derived] Ofili EO, Zappe DH, Purkayastha D, Samuel R, Sowers JR. Antihypertensive and metabolic effects of Angiotensin receptor blocker/diuretic combination therapy in obese, hypertensive African American and white patients. Am J Ther. 2013 Jan;20(1):2-12. doi: 10.1097/MJT.0b013e318230ae66. PMID 22248871
- [Derived] Sowers JR, Raij L, Jialal I, Egan BM, Ofili EO, Samuel R, Zappe DH, Purkayastha D, Deedwania PC. Angiotensin receptor blocker/diuretic combination preserves insulin responses in obese hypertensives. J Hypertens. 2010 Aug;28(8):1761-9. doi: 10.1097/HJH.0b013e32833af380. PMID 20498618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Started | 206 | 206
Completed | 170 | 178
Not Completed | 36 | 28
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Adverse Event | 6 | 4
Not completed — Lost to Follow-up | 5 | 6
Not completed — Protocol Violation | 6 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Abnormal Lab Values | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine | Total
Number analyzed (Participants) | 206 | 206 | 412
Age, Customized [Number; unit: participants]
  < 65 years | 172 (83.5) | 180 (87.4) | 352 (85.4)
  >=65 years | 34 (16.5) | 26 (12.6) | 60 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 148 | 272
  Male | 82 | 58 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP)
Time Frame: Baseline to Week 8
Population: Intent to Treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
mm Hg
  Baseline | 159.7 (7.81) | 159.0 (7.62)
  Week 8 | 131.2 (16.26) | 137.5 (13.52)
  Change from baseline | -28.6 (15.61) | -21.5 (12.58)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP)
Time Frame: Baseline to Weeks 4, 8, 12 and 16
Population: Intent to Treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
mm Hg
  Baseline | 94.9 (7.94) | 93.6 (8.18)
  Week 4 | 85.7 (9.38) | 87.6 (9.20)
  Week 8 | 81.9 (9.87) | 85.1 (8.54)
  Week 12 | 81.1 (9.14) | 82.8 (8.75)
  Week 16 | 80.8 (10.14) | 80.9 (8.66)
  Change from baseline to week 16 | -14.0 (9.90) | -12.7 (8.35)

3. Secondary Outcome: Number of Patients Achieving Blood Pressure (BP) Control by Visit (< 140/90 mm Hg)
Description: Mean sitting systolic blood pressure/mean sitting diastolic blood pressure < 140/90 mm Hg
Time Frame: Weeks 4, 8, 12 16 and End of Study (for patients that did not complete the last visit at week 16)
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
participants
  Week 4 | 91 | 69
  Week 8 | 123 | 102
  Week 12 | 122 | 112
  Week 16 | 124 | 140
  End of study | 133 | 146

4. Secondary Outcome: Number of Patients Achieving Blood Pressure (BP)Control by Visit (< 130/80 mm Hg)
Description: Mean sitting systolic blood pressure/mean sitting diastolic blood pressure < 130/80 mm Hg
Time Frame: Week 4, 8, 12, 16, End of Study (for patients that did not complete the last visit at week 16)
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
participants
  Week 4 | 33 | 18
  Week 8 | 59 | 23
  Week 12 | 57 | 46
  Week 16 | 62 | 65
  End of Study | 68 | 68

5. Secondary Outcome: Change From Baseline in Postprandial Glucose
Description: After a 75 gram anhydrous glucose challenge 2 hours after an oral glucose tolerance test
Time Frame: Week 16
Population: Only those patients who completed the study through week 16 were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
mg/dL
  Baseline visit (0 minutes) | 98.0 (15.91) | 99.4 (19.12)
  Week 16 (0 minutes) | 98.1 (15.68) | 102.8 (17.81)
  Change from baseline to week 16 (0 minutes) | -0.5 (13.71) | 3.4 (18.28)
  Baseline visit (120 minutes) | 123.9 (47.18) | 127.7 (40.30)
  Week 16 (120 minutes) | 126.3 (49.52) | 146.5 (56.51)
  Change from baseline to week 16 (120 minutes) | 2.1 (38.21) | 18.9 (40.88)

6. Secondary Outcome: Change From Baseline in Postprandial Insulin
Description: After a 75 gram anhydrous glucose challenge 2 hours after an oral glucose tolerance test
Time Frame: Week 16
Population: Only those patients who completed the study through week 16 were included in this analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
mg/dL
  Baseline visit (0 minutes) | 19.66 (20.435) | 20.37 (20.583)
  Week 16 (0 minutes) | 23.45 (26.039) | 23.62 (19.267)
  Change from baseline to week 16 (0 minutes) | 3.41 (28.427) | 3.67 (19.170)
  Baseline visit (120 minutes) | 92.04 (82.183) | 95.95 (76.483)
  Week 16 (120 minutes) | 116.04 (129.880) | 120.01 (100.302)
  Change from baseline to week 16 (120 minute) | 24.68 (90.094) | 28.07 (71.674)

7. Secondary Outcome: Change From Baseline in Postprandial Non-esterified Fatty Acids
Description: After a 75 gram anhydrous glucose challenge 2 hours after an oral glucose tolerance test
Time Frame: Week 16
Population: Only those patients who completed the study through week 16 were included in this analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Valsartan/HCTZ (Hydrochlorothiazide) | HCTZ +Amlodipine
Number analyzed (Participants) | 197 | 204
mg/dL
  Baseline visit (0 minutes) | 0.45 (0.208) | 0.47 (0.318)
  Week 16 (0 minutes) | 0.46 (0.194) | 0.47 (0.196)
  Change from baseline to week 16 (0 minutes) | 0.01 (0.249) | 0.00 (0.341)
  Baseline visit (120 minutes) | 0.11 (0.090) | 0.10 (0.116)
  Week 16 (120 minutes) | 0.10 (0.093) | 0.10 (0.056)
  Change from baseline to week 16 (120 minutes) | -0.01 (0.117) | -0.01 (0.120)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other